CLINICAL TRIAL: NCT05944471
Title: The Effect of Breastfeeding Support Provided to Mothers With Insufficient Milk Perception by Telehealth Application on Mothers' Feeding Exclusive Breastfeeding to Their Babies in the First 6 Months
Brief Title: The Effect of Telehealth on Feeding Exclusive Breastfeeding in the Perception of Insufficient Milk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karadeniz Technical University (Other)
Responsible Party: Principal Investigator, Nadire YILDIZ ÇİLTAŞ, Research Assistant, Erzincan Binali Yildirim Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: NYILDIZCILTAS
Record Dates: First submitted 2023-07-06; First posted 2023-07-13 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Breast Feeding; Exclusive Breastfeeding
Keywords: Telehealth; Exclusive Breastfeeding; Self-efficacy
MeSH Terms: conditions — Breast Feeding | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: randomized controlled experimental
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The Inadequate Milk Perception Scale was administered to the mothers to determine the mothers who thought that their milk was inadequate by face-to-face interview method before discharge from the hospital after delivery. Mothers with low scale scores were randomly assigned to the control group as described in the intervention group. Then, Personal Information Form-1, Tendency to Discontinue Breastfeeding Scale and Breastfeeding Self-Efficacy Scale were applied to the mothers. The mothers determined as the control group were called by the investigators via telehealth application between the 2nd-5th days, 13th-17th days, 38th-40th days, 2nd-3rd months, 4th-5th months and at the end of the 6th month and the relevant forms were applied again. No intervention was made to the mothers in the control group.
- Intervention Group (Experimental): Insufficient Milk Perception Scale, Personal Information Form, Tendency to Discontinue Breastfeeding Scale and Breastfeeding Self-Efficacy Scale were also administered to the mothers. After discharge, training videos and written documents were sent to the mothers individually via telehealth application once a week. Visualised messages explaining breastfeeding and that breastmilk is sufficient for the baby were also sent via telehealth application five days a week. Mothers were video-called between 10.00-17.00 on weekdays and live support was provided by the investigators. Mothers in the intervention group were called via telehealth application between the 2nd-5th days, 13th-17th days, 38th-40th days, 2nd-3rd months, 4th-5th months and at the end of the 6th month postpartum and the relevant forms were applied again. In addition, the qualitative questions in the "Semi-structured Interview Form" were asked at the end of the 6th month.
  Interventions: Other: Providing breastfeeding support with Telehealth

INTERVENTIONS:
Other: Providing breastfeeding support with Telehealth — After discharge, training videos on the importance of breast milk and breastfeeding prepared in line with the literature and explained by experts, and written documents (e-brochure, plain text version of breastfeeding trainings) were sent to individual mothers once a week between 10.00-14.00 hours via telehealth application. At the same time intervals, visualised messages explaining breastfeeding and that breast milk is sufficient for the baby were sent via telehealth application five days a week. In addition, if the mothers requested at 10.00-17.00 on weekdays, they were given live support by the researcher for the issues they were curious about breastfeeding by calling the researcher via telehealth application.
  Arms: Intervention Group

SUMMARY:
The goal of this [type of study: The study, which was carried out within the framework of mixed method, is a research using an explanatory sequential design, and its quantitative dimension is a randomized controlled experimental design] is to [The aim of this study is to determine the effect of breastfeeding support given to mothers with inadequate milk perception through telehealth application on mothers' giving only breast milk to their babies for the first six months] in [consisting of primiparous mothers, mothers who had normal vaginal deliveries and mothers with perceived inadequate milk, healthy term babies]. The main question[s] it aims to answer are:

* [What are the experiences of mothers with insufficient milk perception about the breastfeeding support given to their babies with telehealth application and their mothers' experiences about giving only breast milk to their babies for the first six months? ]
* [What is the satisfaction status of mothers with insufficient milk perception towards the breastfeeding support provided by telehealth application? ] Hypotheses of the Study
* [H0: Breastfeeding support provided to mothers with insufficient milk perception through telehealth application has no effect on the mother's exclusive breastfeeding in the first six months. ]
* [H1: Breastfeeding support provided to mothers with insufficient milk perception through telehealth application has an effect on the mother's exclusive breastfeeding for the first six months.]
* [H2: There is a difference between the mean breastfeeding self-efficacy and breastfeeding cessation tendency scale scores of the mothers in the control group and the intervention group with insufficient milk perception.]
* [H3: Mothers have a high level of satisfaction with the breastfeeding support provided by telehealth application.]

Intervention Group: The Inadequate Milk Perception Scale was applied to determine the mothers who thought that their milk was inadequate by face-to-face interview method before discharge from the hospital after delivery. Mothers with low scale scores were assigned to the control group in the first set and to the intervention group in the second set with the help of Research Randomiser (https://www.randomizer.org/). Then, Personal Information Form-1, Tendency to Discontinue Breastfeeding Scale, and Breastfeeding Self-Efficacy Scale were applied to the mothers. After discharge, training videos on the importance of breast milk and breastfeeding and written documents (e-brochure, prose version of breastfeeding trainings) prepared in line with the literature and explained by experts in accordance with the puerperium week between 10.00-14.00 hours were sent to the mothers individually with telehealth application once a week. At the same time intervals, visualised messages explaining breastfeeding and that breast milk is sufficient for the baby were sent via telehealth application five days a week. In addition, if the mothers requested at 10.00-17.00 on weekdays, they were given live support by the researcher for the issues they were curious about breastfeeding by calling the researcher via telehealth application. The mothers in the intervention group were called via telehealth application between the 2nd-5th postpartum days, 13th-17th days, 38th-40th days, 2nd-3rd months, 4th-5th months and at the end of the 6th month and the relevant forms were applied again (at the time period convenient for the mother).

Control Group: The Inadequate Milk Perception Scale was administered to the mothers to determine the mothers who thought that their milk was inadequate by face-to-face interview method before discharge from the hospital after delivery. Then, Personal Information Form-1, Tendency to Discontinue Breastfeeding Scale and Breastfeeding Self-Efficacy Scale were applied to the mothers. The mothers determined as the control group were called by the researcher via telehealth application between the 2nd-5th postpartum days, 13th-17th days, 38th-40th days, 2nd-3rd months, 4th-5th months and at the end of the 6th month by telehealth application and the relevant forms were applied again (at the time period convenient for the mother). No intervention was made to the mothers in the control group, and the woman benefited from routine outpatient clinic services if she requested.

ELIGIBILITY:
* To be able to read and write Turkish and not to have any disability in speaking,
* No desire to breastfeed your baby
* The mother should not have any health problem that would prevent breastfeeding and the baby should not have any health problem that would prevent breastfeeding,
* Having a smartphone and actively using one of the applications such as WhatsApp, Telegram, BIP etc,
* No internet connection problems,
* 37> weeks of gestation,
* Having a baby weighing at least 2500 g,
* Over 18 years of age,
* Primiparous
* Give birth to one healthy baby,
* Vaginal birth

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — primiparous mothers
Enrollment: 70 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
reduce/eliminate the perception of insufficient milk | 1-2 month
  perceiving that mothers who experience inadequate milk perception are able to produce enough milk for their babies

SECONDARY OUTCOMES:
Mothers' Feeding Exclusive Breastfeeding to Their Babies in the First 6 Months | 1-6 month
  to ensure that mothers feed their babies exclusively with breast milk for the first 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No